CLINICAL TRIAL: NCT00595049
Title: Open Label, Non Comparative Study to Investigate the Effect of Bosentan on Pulmonary Artery Remodelling in Pulmonary Arterial Hypertension (PAH).
Brief Title: Pulmonary Artery Remodelling With Bosentan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-416
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hypertension, Pulmonary
Keywords: pulmonary; arterial; artery; hypertension; systemic; sclerosis; scleroderma; remodelling; bosentan; tracleer; intravascular
MeSH Terms: conditions — Hypertension, Pulmonary; Hypertension; Sclerosis; Scleroderma, Diffuse | interventions — Bosentan

ARMS (1):
- bosentan (Experimental)
  Interventions: Drug: bosentan

INTERVENTIONS:
Drug: bosentan — Bosentan 62.5 mg bid for 4 weeks, then 125 mg bid
  Other Names: Tracleer

SUMMARY:
The main purpose of this study is to investigate whether bosentan (Tracleer®) affects the wall thickness of the pulmonary arteries in patients with idiopathic pulmonary arterial hypertension (iPAH) and PAH related to systemic sclerosis (PAH-SSc).

The second purpose is to investigate if bosentan affects the enlargement of small vessels in the lungs in response to natural chemicals in patients with iPAH and PAH-SSc.

ELIGIBILITY:
Inclusion Criteria : · Men or women >18 years of age.·

* Symptomatic (modified NYHA class III) iPAH or PAH-SSc·
* PAH confirmed by right heart catheterization performed within 3 months before enrolment mPAP > 25 mmHg, PCWP < 15 mmHg and PVR > 3 mmHg/l/min.
* Women of childbearing potential must have a negative pre-treatment pregnancy test and use a reliable method of contraception during study treatment and for 3 months after study treatment termination.
* Bosentan naïve patients

Exclusion Criteria : · PAH other than iPAH or PAH-SSc

* Significant vasoreactivity during right heart catheterization defined as a fall in mPAP to < 40 mmHg with a decrease >= 10 mmHg and with a normal cardiac index (>= 2.5 l/min.m2)· Severe obstructive lung disease: FEV1/FVC < 0.5
* Severe restrictive lung disease: TLC < 0.7 of normal predicted value
* Hemoglobin <75% of the lower limit of the normal range· Systolic blood pressure < 85 mmHg
* Body weight < 40 kg
* Pregnancy or breast-feeding
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
* Baseline aminotransferases, i.e., aspartate aminotransferases (AST) and/or alanine aminotransferases (ALT) > 3 times the upper limit of the normal (ULN) range.
* Treatment for iPAH or PAH-SSc within 1 month before start of study treatment, excluding warfarin and acute administration of vasodilators for vascular reactivity testing during heart catheterization.
* Treatment with epoprostenol or other prostacyclin analogs for iPAH or PAH-SSc within 1 month before start of study treatment
* Treatment with glibenclamide (glyburide), fluconazole ketoconazole or ritonavir within 1 week before start of study treatment.
* Current treatment with cyclosporine A or tacrolimus
* Hypersensitivity to bosentan or any of the excipients of its formulation.
* Patient who received an investigational drug (such as sildenafil) within 3 months before start of study treatment
* Conditions that prevent compliance with the protocol or adherence to therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline (BL) to 6 mths in the IVUS-derived measurement of pulmonary artery wall thickness. | Baseline to 6 months
Change from BL to 6 mths in pulmonary microvascular circulation dilator responses to actylcholine (Ach). | Baseline to 6 months

SECONDARY OUTCOMES:
Change from BL to 6 mths in each of the IVUS derived pulmonary artery parameters. | Baseline to 6 months
Change from BL to 6 mths in pulmonary microvascular circulation dilator responses to sodium nitroprusside. | Baseline to 6 months
Correlation between the change from BL to 6 mths of each of the IVUS-derived parameters and the pulmonary microvascular circulation (PMVC) dilator responses versus changes in PVR. | Baseline to 6 months
Correlation between the change from BL to 6 mths of each of the IVUS-derived parameters and the PMVC dilator responses versus changes in 6MWD. | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Celermajer, Professor, Principal Investigator — Royal Prince Alfred Hospital, Camperdown